CLINICAL TRIAL: NCT02013180
Title: Zinc/PSA Ratio as a Novel Biomarker for Prostate Cancer Detection
Status: Completed | Type: Observational
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Mustafa Zafer Temiz, resident, Bagcilar Training and Research Hospital
Other Study IDs: Zinc/PSA
Record Dates: First submitted 2013-12-01; First posted 2013-12-17 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2017-11

CONDITIONS: Prostate Cancer Detection
Keywords: Prostate cancer, PSA, zinc, zinc/PSA
MeSH Terms: conditions — Prostatic Neoplasms; Salivary Gland Adenoma, Pleomorphic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, prostatic tissue

GROUPS / COHORTS (2):
- prostate cancer: prostate adenocarcinoma in pathologic evaluation
- control: benign prostatic diseases in pathologic evaluation

SUMMARY:
Although Prostate Specific Antigen (PSA) is a useful marker for early detection of the prostate cancer, its specivity is not sufficient. Several PSA variations were defined in order to increase the specivity of the test, but they aren't much more effective than the PSA alone for detection of disease.

In older studies reported that, serum and prostatic tissue zinc levels decreased in prostat cancer disease.

In our study we aimed to establish the utility of serum zinc, PSA, free PSA/PSA (fPSA/tPSA), zinc/PSA, levels for early detection of the prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

Patients with LUTS and elevated serum PSA levels and/or suspicious rectal examination

Exclusion Criteria:

usage of zinc included drugs, older prostatic operations, older prostatic radiotherapy, older prostatic biopsies, chronic rectal diseases (anal fissure, hemorrhoid, etc..), PIN(prostatic intraepithelial neoplasia) and ASAP(atypical small acinar proliferation) in pathologic evaluation.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient with LUTS(lower urinary tract symptomps) and elevated serum PSA levels/suspicious rectal examination who undergone transrectal ultrasonography guided prostate biopsy
Sampling Method: Non-Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2012-07; Primary Completion 2013-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bagcilar Training and Research Hospital-Depertmant of Urology, Istanbul, Bagcilar, Turkey (Türkiye)

REFERENCES:
- [Derived] Temiz MZ, Cakir OO, Aykan S, Kucuk SH, Tiryakioglu NO, Bilek G, Tunali NE, Kandirali E, Semercioz A. The use of serum zinc to prostate-specific antigen ratio as a biomarker in the prediction of prostate biopsy outcomes. Biomark Med. 2019 Feb;13(2):59-68. doi: 10.2217/bmm-2018-0260. Epub 2019 Jan 23. PMID 30672309

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prostate Cancer | Control
Started | 119 | 361
Completed | 119 | 361
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prostate Cancer | Control | Total
Number analyzed (Participants) | 119 | 361 | 480
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 177 | 215
  >=65 years | 81 | 184 | 265
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.39 (9) | 64.19 (7.53) | 65.23 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 119 | 361 | 480
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Turkey | 119 | 361 | 480

OUTCOME MEASURES:

1. Primary Outcome: Assesment of Serum Zinc/PSA Ratio in Patients With Prostate Cancer and Benign Prostatic Diseases
Description: Does the zinc/PSA ratio show statistically signifacant difference in patients with prostate cancer?
Time Frame: measurement of serum zinc and PSA levels are performed prior to transrectal prostat biopsy; pathologic evaluation of biopsy specimens are performed within 2-3 weeks
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Prostate Cancer | Control
Number analyzed (Participants) | 119 | 361
ratio | 150.8 [51.8 to 264.1] | 239.6 [145.1 to 357.7]

ADVERSE EVENTS:
Time Frame: 4 years
Description: Not diiferent from the clinicaltrials.gov Definitions
Arm/Group | Prostate Cancer | Control
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/361
Serious Adverse Events (participants affected / at risk) | 0/119 | 0/361
Other Adverse Events (participants affected / at risk) | 0/119 | 0/361

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No